CLINICAL TRIAL: NCT03882320
Title: Medico-economic Evaluation of Sublingual PCA (Zalviso) Versus Oxycodone-PCA in the Management of Postoperative Pain. ''MEZO''
Brief Title: Medico-economic Evaluation of Sublingual PCA (Zalviso) Versus Oxycodone-PCA in the Management of Postoperative Pain.
Acronym: MEZO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Pitié-Salpêtrière Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2018_843_0044
Record Dates: First submitted 2019-03-15; First posted 2019-03-20 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Analgesia
Keywords: Sublingual Patient Controlled Analgesia (PCA); Intravenous Patient Controlled Analgesia (PCA); Patient Controlled Analgesia (PCA)
MeSH Terms: conditions — Agnosia | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sublingual Patient Controlled Analgesia (PCA) (Experimental): Sufentanil Sublingual Patient Controlled Analgesia (PCA)
  Interventions: Procedure: Patient Controlled Analgesia (PCA)
- Intravenous Patient Controlled Analgesia (PCA) (Active Comparator): Oxycodone Intravenous Patient Controlled Analgesia (PCA)
  Interventions: Procedure: Patient Controlled Analgesia (PCA)

INTERVENTIONS:
Procedure: Patient Controlled Analgesia (PCA) — Patient Controlled Analgesia (PCA)

SUMMARY:
More than 230 million surgical operations are been realized all over the world every year. A surgical intervention can cause postoperative acute pain. The management of postoperative acute pain is multimodal and the use of patient-controlled analgesia (PCA) is often a part of this Pain-Management.

Intravenous PCA has established itself as a therapeutic concept and constitutes the reference treatment for the management of postoperative acute pain for the first 48 hours. The PCA offers patients autonomy in managing their pain with the intravenous delivery of morphine on demand.

Since 2017 PCA Zalviso is marketed. It allows the sublingual administration of sufentanil and it does not require venous access. It seems interesting to allow the early rehabilitation of patients who are no longer limited in their movements by an infusion. However, its acquisition cost appears to be higher than that of the intravenous PCA. In order to verify this hypothesis, the investigators propose to compare the set of costs associated with the use of sublingual PCA with those of intravenous PCA in the management of acute postoperative pain (less than 72 hours) in the context of patients benefiting from the placement of a total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* adults
* patients able to express consent
* signed written informed consent form
* patient covered by national health insurance
* patient undergoing total knee arthroplasty and requiring postoperative analgesia with the use of a PCA (patient controlled analgesia)

Exclusion Criteria:

* minors
* obstruction to participate
* patient non covered by national health insurance
* patient requiring a stay in intensive care immediately after the surgery
* patient unable to use a PCA a assessed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Costs of each Intravenous Patient Controlled Analgesia (PCA) | until 72 hours after knee arthroplasty
  Comparison of costs associated with the use of sublingual PCA to those of intravenous PCA

SECONDARY OUTCOMES:
Length of hospitalization | until 72 hours after knee arthroplasty
  Length of hospitalization
Efficiency of acute postoperative pain management | until 72 hours after knee arthroplasty
  Pain intensity is measured with numeric score (scale 0 to 10) (10 is the highest pain intensity; 0 is the score for the absence of pain).
Global satisfaction of the patient | until 72 hours after knee arthroplasty
  Global satisfaction of the patient is measured with " Echelle Visuelle Analogique" EVA score (scale 0 to 10; score 0= no pain; score 10 = pain with the highest intensity)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre NTOUBA, MD, Principal Investigator — CHU Amiens; Sandrine THOMAS SORIOT, MD, Principal Investigator — CHU Amiens; Pierre CORIAT, Pr, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No